CLINICAL TRIAL: NCT06444022
Title: Clinical Study of hAESCs on Prevention of Acute Graft-versus-host Disease After Hematopoietic Stem Cell Transplantation
Brief Title: hAESCs Prevent Acute Graft-versus-host Disease After Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-2019-128
Record Dates: First submitted 2022-07-08; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Acute Graft Versus Host Disease
Keywords: hAESCs

STUDY DESIGN:
Intervention Model Description: The study plans to recruit 18 participants who meet the criteria and is divided into two groups with 9 subjects individually. Infusion of hAESCs/placebo at the day before HSCT and 7th days after HSCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hAESCs (Experimental): Intravenous infusion of hAESCs to 9 subjects at the day before HSCT and 7th days after HSCT. The dose is 1×10^6 cell/kg.
  Interventions: Biological: Human amniotic epithelial stem cells（hAESCs）
- placebo (cell preservation solution) (Placebo Comparator): Intravenous infusion of placebo (cell preservation solution with no hAESCs) to other 9 subjects at the day before HSCT and 7th days after HSCT.
  Interventions: Biological: placebo (cell preservation solution)

INTERVENTIONS:
Biological: Human amniotic epithelial stem cells（hAESCs） — Human Amniotic Epithelial Cells Prevent Acute Graft-versus-host Disease After Hematopoietic Stem Cell Transplantation (hAECs-GVHD)
  Arms: hAESCs
Biological: placebo (cell preservation solution) — Same dose placebo (cell preservation solution) injections as control group
  Arms: placebo (cell preservation solution)

SUMMARY:
This is a parallel controlled clinical study evaluating the safety and efficacy of hAECs in preventing aGVHD after HSCT.

DETAILED DESCRIPTION:
This study is a controlled trial, with 18 subjects enrolled in the experimental group or the control group. The study will consist of four phases, including screening phase, preparation phase, hAESCs treatment phase and observational follow-up period. The cell dose of the experimental group was 1x10^6 cells/kg and the control group is infused placebo (the composition was the same as hAESCs injection excipients, but did not contain hAESCs). The infusion of hAESCs/placebo at the day before HSCT and 7th days after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Standard risk GVHD patients with hematological malignancies older than 18 years;
* High risk GVHD patients with hematological malignancies: haplotype hematopoietic stem cell transplantation patients, donor is female or more than 30 years old;
* Well informed about this study and signed a consent form before the trial;
* Left ventricular ejection fraction (LVEF) ≧ 50%, no evidence of pericardial effusion;
* No evidence of lung infection by X-rays examination;
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1, Hematopoietic cell transplantation - specific comorbidity index (HCT-CI) of 0, 1, 2;
* Normal liver and kidney function: Serum bilirubin≤35µmol/L, AST/ALT was less than 2 times the upper limit of normal value, and serum creatinine ≤130µmol/L

Exclusion Criteria:

* Reduce pretreatment dose or secondary transplantation;
* Participate other clinical trials within 2 months before this study;
* Female, 1) pregnant/nursing period, or 2) have a pregnancy plan during the study period, or 3) have fertility and cannot take effective contraception;
* History of severe allergic disease or is allergic to one or more drugs;
* Patients who are considered unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Follow up closely after intravenous hAESCs therapy to monitor Adverse Event/Serious Adverse Event(AE/SAE) | 1 year
  AE occurring throughout the study period will be evaluated using the CTCAE V5.0 standard. AE/SAE and AESI were evaluated after first hAESCs infusion by laboratory examination, measurement of vital signs, physical examination, and subjects' symptoms to detect new abnormalities and/or deterioration of previous conditions and evaluate the safety of the study.
  hAESCs intravenous infusion is followed up and monitored closely, mainly including vital signs, physical examination, ECOG, electrocardiogram, blood biochemistry, blood RT, urine RT, coagulation laboratory test, imaging examination, type, frequency and severity of AE.

SECONDARY OUTCOMES:
Rate of acute graft-versus-host disease in patients | 1 year
  Occurrence and severity (grade) of Graft-versus-host disease after hAECs infusion
Immune reconstitution 6 months before and after hematopoietic stem cell transplantation | 6 months
  10 days(d) before hematopoietic stem cell transplantation and 1d, 7d±2, 14d±2, 21d±2, 28d±2, 3 month(m) ± 2 days , 6 m ± 2 days, testing expression of immune cells
Hematopoietic stem cell transplantation was performed 10 days before and 1 d, 7 d ±2, 14 d ±2, 21 d±2, 28 d ±2 after transplantation The amount of cytokines in plasma was measured | 1 month
  The amount of cytokines in plasma was measured: TGF-b
Incidence of CMV and EBV infection | 1 year
  Hematopoietic stem cell transplantation after 7 days ±2, 14 days ±2, 21 days±2, 28d±2, 2M±2 days, 3M±2 days, 6M±2 days, 12M±2 days;

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Study Chair — Nanfang Hospital, Southern Medical University